CLINICAL TRIAL: NCT03546751
Title: Extracellular Micro RNA (miR) (Extracellular Vesicle (EV)-Associated & Non-EV-associated miRs) Identify and Mediate Endothelial Dysfunction in Obesity and Obstructive Sleep Apnea in Adolescents & Young Adults
Brief Title: Extracellular microRNA: Biomarkers of Endothelial Dysfunction in Obese Adolescents & Adults With Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Rakesh Bhattacharjee, Associate Professor of Clinical Pediatrics, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 170408
Record Dates: First submitted 2018-05-21; First posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: Endothelial Dysfunction; Micro RNA
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure; Diet; Exercise

STUDY DESIGN:
Intervention Model Description: Comparative Effectiveness Trial
Who Masked: Outcomes Assessor
Masking Description: Investigators will randomize two groups of patients with OSA to receive either CPAP or intensive exercise. The study biostatistician will ensure that matching results in equal distributions of patients based on sex, age, race, severity of OSA, and obesity status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP (Experimental): This arm will consist of patients with obstructive sleep apnea who will be asked to use CPAP nightly to treat their OSA for six months
  Interventions: Device: Continuous Positive Airway Pressure
- Diet and Exercise (Active Comparator): This arm will consist of patients with obstructive sleep apnea who will be asked to engage in dietary management and regular exercise for six months.
  Interventions: Other: Diet And Exercise

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — This device delivers air pressure non invasively through a mask to stent open the upper airway to prevent obstruction during sleep. This is an FDA approved device that has been used for several decades to treat OSA.
  Other Names: CPAP
  Arms: CPAP
Other: Diet And Exercise — This will consist of weekly telephone and monthly face to face visits to monitor and suggest measures to improve diet and regular exercise as conducted by a registered dietician.
  Arms: Diet and Exercise

SUMMARY:
Using a prospective observational approach and a clinical trial design comparing the effectiveness of continuous positive airway pressure to diet and exercise, investigators plan to evaluate how obstructive sleep apnea (OSA) leads to endothelial dysfunction in adolescents and young adults and whether treatment of OSA can improve endothelial dysfunction. Concurrently, investigators will measure miR 92a/miR 210 levels in all subjects at baseline and following therapy to determine whether miR 92a/miR 210 levels reliably predict endothelial dysfunction in patients and responses to therapy.

DETAILED DESCRIPTION:
Investigators will randomize 100 OSA patients (age 13-21) to receive either continuous positive airway pressure (CPAP) plus baseline diet/exercise (n=50) or medical management (intensive diet and exercise; n=50). Only children in whom adenotonsillectomy is contraindicated (morbid obesity, history of adenotonsillectomy, lack of adenotonsillar hypertrophy) will be included. Investigators will conduct a randomized prospective comparative effectiveness study to assess the impact of treatment on OSA on endothelial function (peripheral arterial tonometry-EndoPAT). In addition to diagnostic polysomnography and EndoPAT at baseline, EV (extracellular vesicle) and non EV derived miR 92a/miR 210 concentrations, inflammatory cytokines concentrations, and body anthropometry will be measured. Following 3 mos of therapy and after 6mos of therapy, investigators will re-evaluate EndoPAT, EV and non EV derived miR 92a/miR 210 concentrations, inflammatory cytokines, and body anthropometry.

Throughout the study, investigators will maintain weekly telephone contact and monthly face-to-face visits as per standard of care in both groups to ensure ongoing success. In the medical management group (intensive diet and exercise), diet and exercise will be tracked by maintaining weekly telephone contact and monthly face-to-face visits with a registered dietician. For the CPAP group, investigators will also maintain weekly telephone contact and monthly face-to-face visits with a sleep technician to review mask fitting, and adherence reports, to optimize adherence to CPAP therapy.

Following completion at six months, polysomnography will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy children and young adults with a diagnosis of obstructive sleep apnea based on polysomnography criteria of an obstructive apnea hypopnea index > 10 events/hr.
* For children a BMI range up to 99.7% and for adults BMI up to 32 kg/m2 is used.

Exclusion Criteria:

* The presence of elevated blood pressure
* The presence of diabetes or pre-diabetes
* The presence of craniofacial anomalies
* The presence of neuromuscular disorders
* The presence of syndromic or defined genetic abnormalities
* Pregnancy
* History of smoking (any smoking within the prior 6 mos or >5 pack years total)
* The presence of infectious disease (e.g. including hepatitis B, C, HIV etc.)
* The presence of collagen vascular disease (e.g. lupus, arthritis, scleroderma, polymyositis, mixed-connective tissue disease, vasculitis etc)
* The presence of hepatic disease (including hepatitis fatty liver or cirrhosis)
* The presence of renal disease (including azotemia or clinical proteinuria)
* The presence of cardiopulmonary disease (e.g. known asthma, cystic fibrosis, congenital heart disease)
* Individuals using medications which could affect sleep or breathing (including hypnotics)
* Individuals using chronic anti-inflammatory therapy
* Individuals with any subjects with acute or chronic illness.
* Individuals using anti-hypertensive therapies
* Children with a a BMI > 99.7%
* Adults with a BMI > 32 kg/m2

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Peripheral Arterial Tonometry - Reactive Hyperemic Index | At baseline.
  EndoPAT
Peripheral Arterial Tonometry - Reactive Hyperemic Index | At three months.
  EndoPAT
Peripheral Arterial Tonometry - Reactive Hyperemic Index | At six months.
  EndoPAT

SECONDARY OUTCOMES:
miRNA 92a and miRNA 210 levels | At baseline.
  Serum and Extracellular Vesicle derived miR 92a and miR 210 levels
miR 92a and miR 210 levels | At three months.
  Serum and Extracellular Vesicle derived miR 92a and miR 210 levels
miR 92a and miR 210 levels | At six months.
  Serum and Extracellular Vesicle derived miR 92a and miR 210 levels

IPD SHARING:
Plan to Share IPD: Yes
Intellectual property and data generated under this project will be administered in accordance with both University and NIH policies, including the NIH Data Sharing Policy and Implementation Guidance of March 5, 2003.
  As a part of this application will involve human subjects, investigators believe that the rights and privacy of people who will participate in the research project must be protected at all times. In case other investigators express interest in working with the data, every effort will be made to provide the data to them free of identifiers. However, such endeavors will have to be individually considered and also approved by the University of California (UC) San Diego Human Research Protection Program before any commitments can be made.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 5 years (during the study period)
Access Criteria: Only investigators that are listed as co-investigators with the UC San Diego Human Research Protection Program

REFERENCES:
- [Background] Bhattacharjee R, Khalyfa A, Khalyfa AA, Mokhlesi B, Kheirandish-Gozal L, Almendros I, Peris E, Malhotra A, Gozal D. Exosomal Cargo Properties, Endothelial Function and Treatment of Obesity Hypoventilation Syndrome: A Proof of Concept Study. J Clin Sleep Med. 2018 May 15;14(5):797-807. doi: 10.5664/jcsm.7110. PMID 29734990